CLINICAL TRIAL: NCT05155280
Title: Serotonin Role on Brain Circuits Involved in Food Avoidance in Anorexia Nervosa : Study of Gaze Control and Multimodal Brain Imaging
Brief Title: Serotonin Role on Brain Circuits Involved in Food Avoidance in Anorexia Nervosa
Acronym: SEVIALANO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor received the following instruction from the ANSM : "The sponsor shall conduct toxicity studies in accordance with the applicable guidelines, in particular " ICH guideline M3 (R2) on non-clinical safety studies for the conduct of human cli
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 20CH240; 2021-000906-10 (EudraCT Number)
Record Dates: First submitted 2021-12-01; First posted 2021-12-13 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Anorexia Nervosa
Keywords: anorexia nervosa; serotonin; PET-MRI; eating disorders
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Pathophysiological comparative study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anorexia Nervosa patients (Experimental): 30 patients with anorexia nervosa = 15 with moderate to high anxiety (STAI YB anxiety (STAI YB > 51) and 15 with low anxiety (STAI YB<51).
  A TOBII eye tracker will be realised at Day 1. PET and MRI scans will be acquired at Day 2.
  Interventions: Other: PET imaging using [11C]DASB radioligand.; Behavioral: Eye Tracker
- Controls (Placebo Comparator): 15 healthy volunteers (control group) and a low level of anxiety trait (< 51) A TOBII eye tracker will be realised at Day 1. PET and MRI scans will be acquired at Day 2.
  Interventions: Other: PET imaging using [11C]DASB radioligand.; Behavioral: Eye Tracker

INTERVENTIONS:
Other: PET imaging using [11C]DASB radioligand. — Subjects will be asked to complete a food choice task in PET/MRI. During the task, PET and MRI scans will be acquired simultaneously. This will allow us to see in real time during food choices the brain activations of the subjects. For imaging we will inject the DASB tracer intravenously. This radio ligand is a tracer that allows us to see the cerebral serotoninergic transmission by positron emission tomography.
Behavioral: Eye Tracker — The second technique used is the eye tracker that will allow us to analyze food avoidance behaviors through the eyes. With a "TOBII" eye tracker we wil be able to follow the gaze of the subjects during the food preference task. It is a non-invasive approach.

SUMMARY:
Serotoninergic activity in brain structures involved in food control and avoidance, such as the basal ganglia, is poorly understood in Anorexia Nervosa.

DETAILED DESCRIPTION:
A simultaneous positron emission tomography (PET)- functional magnetic resonance imaging (fMRI) approach and testing of food preferences and choices will provide further insight into the link between potential abnormalities in serotoninergic transmission and the specific food restriction disorder for Anorexia Nervosa. These Data can pave the way for new therapeutic avenues.

ELIGIBILITY:
Common Criteria for inclusion :

* Signature of written consent
* Subject affiliated or entitled to a social security scheme

Inclusion Criteria: Patients with restrictive anorexia nervosa (30 subjects).

* Anorexia nervosa common features : fear of weight gain, dysmorphophobia, BMI < 17.5 kg/ m², amenorrhea
* Absence of food compulsions and purges
* Subgroup 1 (15 subjects) : STAI Y2 anxiety score > 61
* Subgroup 2 (15 subjects) : STAI Y2 anxiety score < 51

Inclusion criteria - Female control subjects (15 subjects)

* BMI between 18.5 and 25 kg/ m²
* Absence of a psychological profile of eating disorder or other psychiatric disorders.

Exclusion Criteria:

* Subjects with an oral contraception and breastfeeding woman
* Subject with heart failure
* Subject treated during the last three months with neuroleptics, and antiparkinsonian drugs, monoamine oxidase (MAO)-A or monoamine oxidase (MOA)-B inhibitors, tricyclic antidepressants, 5HT reuptake inhibitors, thymo regulators (lithium), antiepileptic dugs, codeine derivatives, morphinics, tramadol-containing products (Topalgic, …),dopaminergic drugs.
* Subjects with suspected pregnancy; Test β human chorionic gonadotropin (HCG) positive prior to examination.
* Subjects for whom MRI is contraindicated (pacemaker, intracerebral clips, prosthesis made of ferromagnetic material or claustrophobia).
* Subjects unable to sign written consent for participation in the study.
* Subject deprived of liberty by a judicial or administrative decision

Ages: 16 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-07-08 (Actual)

PRIMARY OUTCOMES:
difference between the two groups of the study for serotonin binding potential | Day 2
  The difference in serotonin binding potential is measured by PET scan of the brain networks between anorexic and control subjects.

SECONDARY OUTCOMES:
correlation between abnormalities in serotonin binding potential and abnormalities in brain activity in resting state | Day 2
  serotonin binding potential is measured with [11C]DASB PET. abnormalities in brain activity is measured on fMRI. correlation between abnormalities in serotonin binding potential and abnormalities in brain activity is quantified by change in the resting state
correlation between abnormalities in serotonin binding potential and abnormalities in brain activity during the food choice tasks. | Day 2
  serotonin binding potential is measured with [11C]DASB PET. abnormalities in brain activity is measured on fMRI. correlation between abnormalities in serotonin binding potential and abnormalities in brain activity is quantified by change during the food choice tasks.
correlation between anxiety profile and brain activity | Day 2
  brain activity is measured on fMRI and anxiety is measured by the score STAI YB.
  STAI YB > 51 = Moderate to high anxiety STAI YB<51 = Low anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Bogdan GALUSCA, PhD, Principal Investigator — Centre Hospitalier Universitaire de Saint Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No